CLINICAL TRIAL: NCT00862134
Title: A Randomized Phase II, Multi-Center, Open-Label Trial of PR104 and Docetaxel in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Randomized, Multi-center, Open-label, Study of PR104 Versus PR104/Docetaxel in Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis indicated low probability of clinically significant result
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR104-2003; NCT00840021 (obsolete NCT alias)
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Granulocyte Colony-Stimulating Factor

ARMS (2):
- Docetaxel 75 mg/m^2 (Active Comparator): Subjects randomized to the docetaxel arm will be administered 75 mg/m^2, IV, every 21 days (an approved dose and schedule)
  Interventions: Drug: docetaxel
- PR104 + 60 mg/m^2 docetaxel (Experimental): Subjects randomized to the PR104/docetaxel arm will be administered 60 mg/m^2 docetaxel, IV, every 21 days plus 770 mg/m^2 PR104, IV, every 21 days and prophylactic G-CSF.
  Interventions: Drug: PR104; Drug: docetaxel; Drug: Granulocyte colony-stimulating factor

INTERVENTIONS:
Drug: PR104 — 770 mg/m^2, IV, every 21 days. Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: PR104 + 60 mg/m^2 docetaxel
Drug: docetaxel — 75 mg/m^2, IV, every 21 days. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Taxotere
  Arms: Docetaxel 75 mg/m^2
Drug: docetaxel — 60 mg/m^2, IV, every 21 days. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Taxotere
  Arms: PR104 + 60 mg/m^2 docetaxel
Drug: Granulocyte colony-stimulating factor — Subjects randomized to PR104/docetaxel will receive prophylactic G-CSF per package insert administration recommendations. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: G-CSF; GCSF
  Arms: PR104 + 60 mg/m^2 docetaxel

SUMMARY:
The current understanding of PR104 justifies the evaluation of PR104 with docetaxel in subjects with Non Small Cell Lung Cancer (NSCLC). These include:

* Aldo-keto reductase 1C3 (AKR1C3). NSCLC has been shown to express high levels of AKR1C3 in about one half of tumors tested. Subjects with high levels of AKR1C3 should have increased activation of PR104 within their tumor.
* Hypoxia. NSCLC has been demonstrated to be a tumor with hypoxia based on both direct tumor measurements (oxygen electrodes) and hypoxic positron emission tomography (PET) imaging. Tumor hypoxia in NSCLC should be sufficient to activate PR104 to its active metabolites PR104H and PR104M.
* Preclinical data. The use of docetaxel and PR104 alone and in combination in preclinical models demonstrates activity of PR104 as a single agent and supraadditive activity when PR104 and docetaxel are used in combination.
* Manageable toxicity. PR104 and docetaxel with Granulocyte Colony-stimulating Factor (G-CSF) have been combined in a prior phase I study. A Maximum Tolerated Dose (MTD) has been identified and the major toxicities of this combination are understood.

The current study will provide an estimate of the activity of PR104 in subjects with NSCLC. This information will prove valuable in defining the future clinical development of PR104, and in determining if PR104 has sufficient activity in NSCLC to warrant a larger phase III registration study in this indication.

Primary objectives

• Estimate the response rate (RR) of PR104/docetaxel

Secondary objectives

* Evaluate survival
* Evaluate progression free survival (PFS)
* Evaluate time to progression (TTP)
* Evaluate safety
* Evaluate the pharmacokinetics of PR104 and its metabolites
* Evaluate the pharmacokinetics of docetaxel
* Evaluate the tumor hypoxia using 18F-fluoromisonidazole (18F-MISO) PET imaging
* Collect diagnostic biopsy samples for the determination of AKR1C3
* Collect plasma samples for assessment of potential biomarkers of tumor hypoxia

DETAILED DESCRIPTION:
A randomized phase II, multi-center, open-label, study of docetaxel versus docetaxel/PR104.

Following informed consent, subjects will undergo baseline evaluation with history, physical exams, blood work and disease assessment. Selected subjects will undergo PET imaging with F18 fluoromisonidazole (F18-FMISO) and Fludeoxyglucose (FDG) for assessment of hypoxia and glucose metabolism, and pharmacokinetics of PR104.

Subjects will be randomized between arm 1 consisting of docetaxel, 75 mg/m^2, administered intravenously (IV), every 21 days (an approved dose and schedule) and arm 2 consisting of docetaxel, 60 mg/m^2 with PR104 at 770 mg/m^2, IV, every 21 days. Subjects randomized to PR104/docetaxel will receive prophylactic G-CSF. One cycle will be 21 days in duration. Subjects will be evaluated weekly. A disease assessment will be performed every six weeks. Subjects with progression will be removed from study. Subjects with a response or stable disease may continue on study if this is considered beneficial by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with locally advanced or metastatic NSCLC (stage IIIb/IV) who have relapsed following adjuvant or first line therapy with a platinum containing regimen, and are appropriate candidates for treatment with single agent docetaxel
* Confirmed NSCLC by prior pathological analysis (tissue aspirate or biopsy)
* At least 21 days from prior chemotherapy
* At least 30 days from prior irradiation therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of 12 weeks or more
* Adequate hematologic function [Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; platelet count ≥100x10^9/L; hemoglobin ≥8.5 g /dL maintained in the absence of red blood cell transfusions; and prothrombin time international normalized ratio ≤1.7; or prothrombin time ≤2 seconds above control)
* Adequate hepatic function (albumin ≥2.8 g/dL; total bilirubin ≤2 mg/dL [51.3 μmol/L]; and alanine aminotransferase and aspartate aminotransferase ≤1.5 times the upper limit of the normal range)
* Adequate renal function (serum creatinine ≤2.0 times the upper limit of the normal range or creatinine clearance ≥60 mL/min).
* At least one untreated target lesion that could be measured in one dimension, according to the Response Evaluation Criteria in Solid Tumors (RECIST)

Exclusion Criteria:

* Previous treatment with docetaxel (prior treatment with paclitaxel permitted)
* Receipt of more than one prior systemic chemotherapy regimen
* Active concomitant malignancy likely to effect any of the primary or secondary outcome measures in the current study
* Women who are pregnant, breast-feeding or planning to become pregnant during the study
* Men or women of reproductive-potential who are unwilling to use an effective method of contraception during the study and for 30 days following the last dose
* Evidence of a significant medical disorder or laboratory finding that, in the opinion of the Investigator, compromises the subject's safety during study participation
* Active Central Nervous System (CNS) metastatic disease requiring intervention
* Less than 4 weeks since major surgery
* Known human immunodeficiency virus (HIV) positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (25):
  - Sharp Clinical Oncology Research, San Diego, California
  - University of Miami/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Orchard Research, LLC, Skokie, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - St. Francis Health Services, Beech Grove, Indiana
  - McFarland Clinic/William R. Bliss Cancer Center, Ames, Iowa
  - Iowa Blood & Cancer Care, Cedar Rapids, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Baton Rouge General/Penington, Baton Rouge, Louisiana
  - Annapolis Oncology Center, Annapolis, Maryland
  - Lapidus Cancer Center/Sinai Hospital, Baltimore, Maryland
  - Kalamazoo Hematology & Oncology, Kalamazoo, Michigan
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - VA Medical Center, Durham, North Carolina
  - Piedmont Hematology Oncology Associates, PLLC, Winston-Salem, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - ACORN, Memphis, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology - Allison Cancer Center, Midland, Texas
  - Scott & White Memorial Hospital, Temple, Texas
- McGill University, Montreal, Quebec, Canada
- Waikato District Health Board, Hamilton, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel: 75 mg/m^2 docetaxel, IV, every 21 days
- PR104 + Docetaxel: Subjects randomized to the PR104/docetaxel arm will be administered 60 mg/m^2 docetaxel, IV, every 21 days plus 770 mg/m^2 PR104, IV, every 21 days and prophylactic Granulocyte Colony-stimulating Factor (G-CSF).
Period: Overall Study
Arm/Group | Docetaxel | PR104 + Docetaxel
Started | 19 | 23
Completed | 8 | 11
Not Completed | 11 | 12
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Sponsor terminated study | 5 | 7
Not completed — Adverse Event | 2 | 2
Not completed — Withdrew prior to dosing | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- PR104 + Docetaxel: Subjects randomized to the PR104/docetaxel arm will be administered 60 mg/m^2 docetaxel, IV, every 21 days plus 770 mg/m^2 PR104, IV, every 21 days and prophylactic G-CSF.
- Total: Total of all reporting groups
Arm/Group | Docetaxel | PR104 + Docetaxel | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 23
  >=65 years | 5 | 14 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (7.78) | 64 (7.58) | 63 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39
  Canada | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved a Response (Complete or Partial) After Receiving PR104/Docetaxel Versus Docetaxel Alone
Description: Defined as the number of subjects with complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) criteria
Time Frame: Participants were followed for the duration on study, an average of 4 months
Measure: Number; unit: participants
Arm/Group | Docetaxel | PR104 + Docetaxel
Number analyzed (Participants) | 17 | 21
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 1 | 3

2. Secondary Outcome: Safety and Tolerability: Serious Adverse Events
Description: The number of participants with at least one Serious Adverse Event was measured.
Time Frame: 30 days following last administration of study treatment
Measure: Number; unit: participants
Arm/Group | Docetaxel | PR104 + Docetaxel
Number analyzed (Participants) | 17 | 23
participants | 8 | 5

3. Secondary Outcome: Positive Aldo-keto Reductase 1C3 (AKR1C3) Expression in Participating Patients
Description: AKR1C3 was evaluated on a semi-quantitative scale, and the percentage of cells staining at each of the following four levels was recorded: 0 (unstained), 1+ (weak staining), 2+ (moderate staining) and 3+ (strong staining).
  Patients with a strong staining score (3+) were considered to be AKR1C3 positive
Time Frame: Within 1 year of enrollment
Measure: Number; unit: participants
Arm/Group | Docetaxel | PR104 + Docetaxel
Number analyzed (Participants) | 11 | 12
participants | 5 | 8

ADVERSE EVENTS:
Arm/Group | Docetaxel | PR104 + Docetaxel
Serious Adverse Events (participants affected / at risk) | 8/17 | 5/23
Other Adverse Events (participants affected / at risk) | 17/17 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=17) | PR104 + Docetaxel (N=23)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Chest Pain (atypical) (General disorders) | 2 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0
Ileus, GI (Gastrointestinal disorders) | 0 | 0
Acute RLL Pneumonia (Infections and infestations) | 2 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Gastrointestinal Bleed (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Gastroenteritis (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Spinal Cord Compression (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=17) | PR104 + Docetaxel (N=23)
Anaemia (Blood and lymphatic system disorders) | 10 | 14
Neutropenia (Blood and lymphatic system disorders) | 10 | 14
Leukopenia (Blood and lymphatic system disorders) | 10 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Fatigue (General disorders) | 9 | 8
Non-cardiac chest pain (General disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Diarrhoea (General disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastric ileus (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Candidiasis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Delirium (Psychiatric disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Hepatitis C virus (Investigations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Single site data may be published/presented prior to the publication of multi-center data from overall study if agreed to by the sponsor in writing, or 12 months have elapsed following termination or completion of the study, whichever comes first.